CLINICAL TRIAL: NCT01640184
Title: Study of the Efficacy and Safety on the Ultrasonic Ablation Treatment for Secondary Hyperthyroidism in Chronic Kidney Disease Patients.
Brief Title: Efficacy and Safety of Ultrasonic Ablation to Treat Secondary Hyperparathyroidism in Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongliang Zhang, MD (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor-Investigator, Dongliang Zhang, MD, associate professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-079; Z121107001012138 (Other Grant/Funding Number: Beijing Municipal Science and Technology Commission); 2001-2002-02 (Other Grant/Funding Number: The capital health research and development of special)
Record Dates: First submitted 2012-07-09; First posted 2012-07-13 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Hyperparathyroidism; Disorders of Parathyroid Gland
Keywords: hyperparathyroidism; vitamin D; ultrasonic ablation; surgery
MeSH Terms: conditions — Hyperparathyroidism; Parathyroid Diseases | interventions — Parathyroidectomy; Oral Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active vitamin D (Active Comparator): Patients in oral medicine group will be treated by active vitamin D and other general treatments according to the suggestions in Kidney Developement Improvement Global Outcomes (KDIGO) guidelines.
  Interventions: Drug: Active vitamin D
- Ultrasonic ablation (Experimental): Patients in Ultrasonic ablation group will be treated by ultrasound guided percutaneous parathyroid gland radio frequency ablation.
  Interventions: Procedure: Ultrasonic ablation
- Parathyroidectomy (Active Comparator): Patients in parathyroidectomy group will be treated by parathyroid surgery.
  Interventions: Procedure: Parathyroidectomy

INTERVENTIONS:
Procedure: Parathyroidectomy — sHPT patients with enlarged glands (≥3)will be randomized into parathyroidectomy group or ultrasonic ablation group. Patients in parathyroidectomy will get parathyroid surgery.
  Other Names: Parathyroid surgery
  Arms: Parathyroidectomy
Drug: Active vitamin D — CKD patients suffered from sHPT with 1-3 enlarged gland(s) and without indication of parathyroidectomy will be randomized to oral medicine therapy group or ultrasonic ablation therapy group. Patients in oral medicine group will be treated by active vitamin D and other general treatments, such as dietary phosphate restriction and phosphate binders, according to the suggestions in KDIGO guidelines.
  Other Names: Oral medicine
  Arms: Active vitamin D
Procedure: Ultrasonic ablation — CKD-sHPT patients with enlarged parathyroid gland(s) randomized into the ultrasonic ablation group will be treated by ultrasound guided percutaneous parathyroid gland radio frequence ablation. According to the indications of parathyroid surgery, the patients will be divided into two sub-groups. The outcomes of these patients will be compared to the oral medicine group and the parathyroidectomy group, respectively.
  Other Names: Ultrasonic intervention
  Arms: Ultrasonic ablation

SUMMARY:
It is difficulty for the treatment of secondary hyperparathyroidism in the chronic kidney disease (CKD) patients who had not succeeded medical therapy and could not get parathyroidectomy. The investigators suppose that ultrasonic ablation may be a valuable alternative treatment that help control secondary hyperparathyroidism in CKD patients presenting with enlarged parathyroid gland(s) visible at ultrasonography.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism (sHPT) is common in patients with chronic kidney disease (CKD), including those who are undergoing long-term dialysis treatments. sHPT is damaged for bone system, blood system, cardiovascular system, and so on. The treatment of the sHPT of CKD's patient includes dietary phosphate restriction, the use of medicines, and parathyroidectomy. In the mainland of China, there are not certain useful medicines to treat sHPT, including the derivatives of vitamin D, calcimimetic agent, non calcium aluminum phosphate binders. Furthermore, medical therapy is not always successful in achieving adequate control of sHPT. Oral medications have efficacy limitations as well as side-effects. Otherwise, surgery treatment can only be used for the patients with enlarged parathyroid gland(s). The patients may suffer from the injury of operation, hypoparathyroidism, or recurrence of hyperparathyroidism after parathyroidectomy.

Then ultrasonic ablation may become a valuable alternative treatment that help control sHPT in selected patients presenting with enlarged parathyroid gland(s) visible at ultrasonography,.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 - 75 years.
* Patients with parathyroid nodular or diffuse hyperplasia demonstrated on ultrasound imaging or radioisotope scan.
* CKD patients in stage 5, with elevated intact parathyroid hormone (iPTH) levels > 800pg/mL.
* CKD patients have been followed up more than 6 months.

Exclusion Criteria:

* Primary or Tertiary Hyperparathyroidism (hyperparathyroidism after kidney transplantation).
* Patient who underwent total parathyroidectomy and without enlarged parathyroid gland(s).
* Known history of parathyroid or other neoplasias in the neck region.
* History of neck irradiation.
* Major surgery of neck in the last 3 months or other major surgery projected in the subsequent 4 months.
* Pregnant or lactating woman.
* Patient receiving drugs such as phenobarbital, phenytoin, rifampicin, sucralfate, steroids, flecainide, thioridazine, or most tricyclic antidepressants which could affect vitamin D metabolism.
* Treatment with vitamin D derivatives, cinacalcet or other calcimimetics within the past 6 months.
* Patients who are currently participating in another clinical trial.
* The expected live time is less than 1 year.
* Patients suffered from acute myocardial infraction, acute congestive heart failure, or stroke in last 6 months.
* Patients whose concurrent illnesses, disability, or geographical residence would hamper attendance at required study visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linxue Qian, Doctor, Principal Investigator — Beijing Friendship Hospital; Dongliang Zhang, Doctor, Study Director — Beijing Friendship Hospital; Wenhu Liu, Doctor, Study Chair — Beijing Friendship Hospital
Locations (2):
- China (2):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Vitamin D: Patients in oral medicine group will be treated by active vitamin D and other general treatments according to the suggestions in KDIGO guidelines.
  Active vitamin D: CKD patients suffered from sHPT with 1-3 enlarged gland(s) and without indication of parathyroidectomy will be randomized to oral medicine therapy group or ultrasonic ablation therapy group. Patients in oral medicine group will be treated by active vitamin D and other general treatments, such as dietary phosphate restriction and phosphate binders, according to the suggestions in KDIGO guidelines.
Period: Overall Study
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy
Started | 34 | 23 | 22
Completed | 26 | 21 | 20
Not Completed | 8 | 2 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy | Total
Number analyzed (Participants) | 34 | 23 | 22 | 79
Age, Continuous [Mean (Full Range); unit: years] | 56.3 [20 to 74] | 52.0 [24 to 73] | 55.2 [26 to 69] | 55.3 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 13 | 45
  Male | 14 | 11 | 9 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 34 | 23 | 22 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 34 | 23 | 22 | 79
Ca-baseline [Mean (Standard Deviation); unit: mmol/L] — Blood level of Calcium on baseline.
  mmol/L | 2.31 (0.27) | 2.43 (0.30) | 2.53 (0.23) | 2.41 (0.30)
P-baseline [Mean (Standard Deviation); unit: mmol/L] — Blood level of phosphorus on baseline.
  mmol/L | 1.95 (0.49) | 2.14 (0.66) | 2.12 (0.45) | 2.10 (0.51)
iPTH-baseline [Mean (Standard Deviation); unit: ng/ml] — Blood level of intact parathyroid hormone on baseline.
  ng/ml | 239.84 (299.01) | 1550.6 (521.7) | 1779.9 (514.1) | 1201.8 (498.7)
BALP-baseline [Mean (Standard Deviation); unit: microgram/L] — Blood level of Bone-alkaline phosphatase (BALP) on baseline.
  microgram/L | 17.31 (6.38) | 18.84 (17.94) | 19.27 (14.87) | 17.98 (13.32)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Achieving the Target on Blood Intact Parathyroid Hormone Level According to Kidney Development Improvement Global Outcome (KDIGO) Guidelines.
Description: The blood levels of intact parathyroid hormone (iPTH) will be detected every 3 months for stable patients. The blood test will be more frequent, at least once per-month, after the ultrasonic ablation treatment, surgery, or during the impulse therapy of active vitamin D with large doses.
Time Frame: 12 months
Population: Number of participants analyzed is the number of patients completed study.
Measure: Number; unit: percentage of participants
Groups:
- Active Vitamin D: Patients in oral medicine group will be treated by active vitamin D and other general treatments according to the suggestions in KDIGO guidelines.
  Active vitamin D: chronic kidney disease (CKD) patients suffered from secondary hyperparathyroidism (sHPT) with 1-3 enlarged gland(s) and without indication of parathyroidectomy will be randomized to oral medicine therapy group or ultrasonic ablation therapy group. Patients in oral medicine group will be treated by active vitamin D and other general treatments, such as dietary phosphate restriction and phosphate binders, according to the suggestions in KDIGO guidelines.
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy
Number analyzed (Participants) | 26 | 21 | 20
percentage of participants | 30.8 | 57.1 | 90.0

2. Secondary Outcome: Incidence of Injury on the Recurrent Laryngeal Nerve (RLN).
Description: Comparison of the incidence of RLN injury between ultrasonic ablation group and parathyroidectomy group.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Ultrasonic Ablation | Parathyroidectomy
Number analyzed (Participants) | 21 | 20
participants | 0 | 2

3. Secondary Outcome: Changes of the Blood Levels on Calcium During 12 Months.
Description: The blood levels of calcium will be detected at least once every 3 months and will be compared to the baseline levels.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy
Number analyzed (Participants) | 26 | 21 | 20
mmol/L | 2.34 (0.22) | 1.84 (0.21) | 1.93 (0.26)

4. Secondary Outcome: Changes of Blood Levels on Phosphorus During 12 Months.
Description: The blood levels of phosphorus will be detected at least once every 3 months and will be compared to the baseline levels.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy
Number analyzed (Participants) | 26 | 21 | 20
mmol/L | 1.91 (0.41) | 1.51 (0.29) | 1.29 (0.33)

5. Secondary Outcome: Changes of Blood Levels on iPTH During 12 Months.
Description: The blood levels of iPTH will be detected at least once every 3 months and will be compared to the baseline levels.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy
Number analyzed (Participants) | 26 | 21 | 20
ng/ml | 252.2 (172.0) | 372.1 (253.6) | 246.5 (228.4)

6. Secondary Outcome: Changes of Blood Levels on Bone Specific Alkaline Phosphatase.
Description: The blood levels of bone specific alkaline phosphatase will be detected at least once every 3 months and will be compared to the baseline levels.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: microgram/L
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy
Number analyzed (Participants) | 26 | 21 | 20
microgram/L | 13.60 (5.86) | 19.48 (17.33) | 19.20 (17.95)

ADVERSE EVENTS:
Arm/Group | Active Vitamin D | Ultrasonic Ablation | Parathyroidectomy
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/34 | 5/23 | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Vitamin D (N=34) | Ultrasonic Ablation (N=23) | Parathyroidectomy (N=22)
Death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — The reason of death was unclear. The patient had been dead when family found.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Vitamin D (N=34) | Ultrasonic Ablation (N=23) | Parathyroidectomy (N=22)
Hypocalcemia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 15 (15) — Blood ionized calcium level decreased caused by surgery.
Hoarse (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 8 (8) — Recurrent laryngeal nerve injury caused by surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No